CLINICAL TRIAL: NCT02428322
Title: Randomized, Double-blind, Placebo Controlled Trial of Vitamin D3 Supplementation on Clinical, and Subjective Symptoms of Paediatric Asthma
Brief Title: Trial of Vitamin D3 Supplementation in Paediatric Asthma
Acronym: NCHVitDAst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conor Kerley (Other)
Responsible Party: Sponsor-Investigator, Conor Kerley, PhD candidate, University of Dublin, Trinity College
Organization: University of Dublin, Trinity College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NCH-ASTHMA-VIT.D
Record Dates: First submitted 2014-10-10; First posted 2015-04-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 2,000iu vitamin D3 per day for 15 weeks
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: VItamin D3
- Placebo (Placebo Comparator): An identical placebo capsule daily for 15 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Soft gel capsules will be identical to the vitamin D intervention but contain no vitamin D.
Dietary Supplement: VItamin D3 — Soft gel capsules will contain 2,000IU vitamin D.
  Arms: Intervention

SUMMARY:
Epidemiological and observational studies have linked vitamin D deficiency with increased asthma/allergy incidence . Vitamin D insufficiency (<75nmol/L) has been associated with increased incidence of severe childhood asthma. Further, high 25(OH)D levels were associated with reduced risk of recent hospitalization, lower use of anti-asthmatic medication and lower airway hyper-responsiveness in childhood asthmatics. The association between vitamin D and allergy and asthma appears to be stronger in children than adults, with some even suggesting that childhood asthma may may be caused by VDD.

DETAILED DESCRIPTION:
Asthmatic children will be recruited in winter. After baseline testing, children will be randomized to take 2,000iu vitamin D or placebo daily for 15 weeks. After the 15 weeks, testing will be repeated. Tests involve blood draws, questionnaires and breathing tests.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of asthma
* Ability to perform pulmonary function tests
* Established on anti-asthmatic pharmacotherapy with no expected change

Exclusion Criteria:

* Use of medications that influence vitamin D metabolism or absorption
* Chronic, non-asthma medical issues e.g. endocrine, hepatic, renal, or bone-disease

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Paediatic Asthma Control Test (P-ACT) | 15 weeks

SECONDARY OUTCOMES:
Global Initiative for Asthma Score | 15 weeks
Pulmonary function | 15 weeks
  FEV1, FVC, FEV1:FVC
Height velocity | 15 weeks
  Rate of change in height
Biochemical markers (25(OH)D, total IgE, total calcium, albumin, PTH, phosphate, hsCRP, IgA and ECP. | 15 weeks
Mini paediatric asthma quality of life questionnaire | 15 weeks
Asthma Diary | 15 weeks
  A 13 item diary to be filled out weekly by parents/gaurdians.

CONTACTS AND LOCATIONS:
Overall Officials: Basil Elnazir, MD, Principal Investigator — National Children's Hospital, Dublin 24, Ireland